CLINICAL TRIAL: NCT05992402
Title: Readiness Brain Operation Optimization Training (ReBOOT) for Epilepsy Surgery
Acronym: ReBOOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kayela Arrotta (Other)
Collaborators: American Psychological Association (APA) (Other); American Epilepsy Society (Other); The Cleveland Clinic (Other)
Responsible Party: Sponsor-Investigator, Kayela Arrotta, Principal Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 23-212
Record Dates: First submitted 2023-07-24; First posted 2023-08-15 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in this arm will receive 2 one-on-one virtual education sessions as well as 4 virtual group education sessions prior to their epilepsy surgery.
  Interventions: Behavioral: ReBOOT program
- Treatment-as-Usual (No Intervention): Treatment as usual but will also receive three brief 5-minute phone calls over 6-weeks after initial enrollment. These phone calls are not therapeutic in nature but provide control participants with brief engagement in study-related activities to ensure that any benefits seen between groups are not simply attributable to study participation.

INTERVENTIONS:
Behavioral: ReBOOT program — This is a virtual cognitive intervention led by a clinical neuropsychologist. Participants will attend 2 one-on-one individual sessions and 4 group sessions prior to their epilepsy surgery. Groups will be made up of 3-10 participants. The intervention is designed to provide participants with information about possible changes and/or challenges they may experience after epilepsy surgery, as well as cognitive strategies to implement prior to surgery to increase effectiveness of compensation for any new cognitive difficulties that may be experienced following surgery.
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to learn if new educational program prior to epilepsy surgery can either decrease the risk of cognitive decline after surgery or be a help to those patients who experience a decline after undergoing epilepsy surgery.

Participants will participate in 2 individual virtual sessions and 4 virtual group sessions over the course of 5-6 weeks prior to their epilepsy surgery. They will asked to fill out online surveys and questionnaires at various times throughout the study, up to 12 months after their surgery.

To see if the educational program works, researchers will compare those participating in the educational program with those that are receiving the standard epilepsy care prior to surgery.

DETAILED DESCRIPTION:
In this prospective, controlled, randomized study, the researchers aim to assess the feasibility and effectiveness of a cognitive intervention in those with epilepsy. They will implement a novel prehabilitation program for patients who have been recommended for epilepsy surgery and will track retention, and adherence to understand the feasibility of the program. Researchers will gather patient data regarding satisfaction with the prehabilitation program and elicit qualitative feedback from patients to further refine the program. To assess intervention efficacy, researchers will compare patients who undergo the prehabilitation program to a treatment-as-usual control group on outcome measures related to quality of life, compensatory strategy use, psychosocial factors, and surgical satisfaction.

The study team will accomplish these objectives by comparing participants that are randomly assigned to the ReBOOT intervention arm (2 individual, virtual sessions and 4 virtual, group sessions over the course of 5-6 weeks) to those participants assigned to the control arm (standard epilepsy care). Researchers will measure the effects and feasibility of the intervention through the use attendance tracking, homework adherence, and health and quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Adults, aged 18-60 years old, with diagnosed epilepsy who have been confirmed as an appropriate surgical candidate by their epileptologist
* Able to independently provide informed consent
* Fluent in English
* Reading abilities at or above 8th grade level as determined by the Wide Range Achievement Test- 4th Edition (WRAT-4), Reading subtest.
* Internet access and the ability to participate in online video streaming
* No history of resective or ablative neurosurgery, but this does not include neuromodulation therapies for epilepsy (e.g., RNS, VNS, DBS)
* Willing and able to participate in cognitive intervention

Exclusion Criteria:

* Any patient that has engaged in any form of cognitive rehabilitation/intervention within the last 6 months
* Ongoing litigation related to the cause of epilepsy, unless litigation is related to short term or long-term disability application.
* Undergoing intensive medical treatment for serious or life-threatening illness (e.g., chemotherapy, etc.) that would impact study participation.
* Serious psychiatric condition that could interfere with participation, such as schizophrenia, active psychosis, active mania, and current suicidal ideation.
* Significant hearing and/or vision loss that would preclude them from participating in remote cognitive testing and engaging in the cognitive intervention.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Intervention attendance | 5-6 Weeks post study enrollment
  As determined by weekly group attendance and the number of weeks it takes each patient to complete all four rotating sessions
Rate of Homework Completion | 5-6 Weeks post study enrollment
  As determined by self-reported whether or not patient attempted to complete or completed their homework
Study Attrition | 5-6 Weeks post study enrollment
  As determined by number of patients who do not complete the ReBOOT program and the reasons why
Intervention Efficacy based on Quality of Life | 5-6 weeks post study enrollment, 6 month, 12 month
  As assessed by the Quality of Life in Epilepsy questionnaire (Min/Max: 0-100, higher score means better outcome)

SECONDARY OUTCOMES:
Change in Subjective Cognitive Function | 5-6 weeks post study enrollment, 6 month, 12 month
  As assessed by the Memory Assessment Clinics Scale for Epilepsy (Min/Max: 30-150, Higher score means better outcome) and the Everyday Compensation Scale (Min/Max: 0-220, higher score means better outcome)
Change in Stress | 5-6 weeks post study enrollment, 6 month, 12 month
  As assessed by the Perceived Stress Scale 4 (Min/Max: 0-16, higher score means worse outcome)
Change in Mood | 5-6 weeks post study enrollment, 6 month, 12 month
  As assessed by the Patient Health Questionnaire (Min/Max: 0-24, higher score means worse outcome) and the Generalized Anxiety Disorder (Min/Max: 0-21, higher score means worse outcome)
Surgery Satisfaction assessed by Epilepsy Surgery Satisfaction Questionnaire | 6 month, 12 month
  Min/Max: 19-133, higher score means better outcome
Intervention Efficacy based on Functional Status | 5-6 weeks post study enrollment, 6 month, 12 month
  As assessed by the Instrumental Activities of Daily Living-Compensation questionnaire (Min/Max: 27-216, higher score means worse outcome)
Satisfaction with ReBOOT | 5-6 weeks post study enrollment
  As assessed by the qualitative Satisfaction of ReBOOT questionnaire and qualitative feedback
Change in Self-Efficacy | 5-6 weeks post study enrollment, 6 month, 12 month
  As assessed by the General Self-Efficacy Scale questionnaire (Min/Max: 10-40, higher score means greater self-efficacy)
Change in Locus of Control | 5-6 weeks post study enrollment, 6 month, 12 month
  As assessed by the Multidimensional Health Locus of Control questionnaire (Min/Max: 24-144, higher score means greater locus of control)
Change in Word List Recall | Pre-surgery and 6 Months Post-surgery
  As assessed by the Rey Auditory Verbal Learning Task (Min/Max: 50-150, Higher score means better outcome).
Change in Story Recall | Pre-surgery and 6 Months Post-surgery
  As assessed by the Wechsler Memory Scale - 4th Edition Logical Memory (Min/Max: 1-19, Higher score means better outcome).
Change in Visual Memory Recall | Pre-surgery and 6 Months Post-surgery
  As assessed by the Wechsler Memory Scale - 4th Edition Visual Reproductions (Min/Max: 1-19, Higher score means better outcome).
Change in Naming | Pre-surgery and 6 Months Post-surgery
  As assessed by the Boston Naming Test (Min/Max: 0-60, Higher score means better outcome).
Change in Attention | Pre-surgery and 6 Months Post-surgery
  As assessed by the Wechsler Adult Intelligence Scale - 4th Edition Digit Span (Min/Max: 1-19, Higher score means better outcome).
Change in Problem Solving | Pre-surgery and 6 Months Post-surgery
  As assessed by the Wisconsin Card Sorting Test (Min/Max: 50-150, Higher score means better outcome).
Change in Mental Flexibility | Pre-surgery and 6 Months Post-surgery
  As assessed by the Trail Making Test Part B (Min/Max: 20-80, Higher score means better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Kayela Arrotta, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu SY, Yang XL, Chen B, Hou Z, An N, Yang MH, Yang H. Clinical outcomes and quality of life following surgical treatment for refractory epilepsy: a systematic review and meta-analysis. Medicine (Baltimore). 2015 Feb;94(6):e500. doi: 10.1097/MD.0000000000000500. PMID 25674741
- [Background] Sherman EM, Wiebe S, Fay-McClymont TB, Tellez-Zenteno J, Metcalfe A, Hernandez-Ronquillo L, Hader WJ, Jette N. Neuropsychological outcomes after epilepsy surgery: systematic review and pooled estimates. Epilepsia. 2011 May;52(5):857-69. doi: 10.1111/j.1528-1167.2011.03022.x. Epub 2011 Mar 22. PMID 21426331
- [Background] Busch RM, Floden DP, Ferguson L, Mahmoud S, Mullane A, Jones S, Jehi L, Bingaman W, Najm IM. Neuropsychological outcome following frontal lobectomy for pharmacoresistant epilepsy in adults. Neurology. 2017 Feb 14;88(7):692-700. doi: 10.1212/WNL.0000000000003611. Epub 2017 Jan 13. PMID 28087827
- [Background] Pauli C, Schwarzbold ML, Diaz AP, de Oliveira Thais MER, Kondageski C, Linhares MN, Guarnieri R, de Lemos Zingano B, Ben J, Nunes JC, Markowitsch HJ, Wolf P, Wiebe S, Lin K, Walz R. Predictors of meaningful improvement in quality of life after temporal lobe epilepsy surgery: A prospective study. Epilepsia. 2017 May;58(5):755-763. doi: 10.1111/epi.13721. Epub 2017 Mar 23. PMID 28332703
- [Background] Qiu Y, Zhang J, Yan Y, Liu W, Zhan S, Huang P, Deng Y. Predictors of meaningful improvement in quality of life after selective amygdalohippocampectomy in Chinese patients with refractory temporal lobe epilepsy: A prospective study. Epilepsy Behav. 2019 Aug;97:1-7. doi: 10.1016/j.yebeh.2019.05.006. Epub 2019 Jun 7. PMID 31181423
- [Background] Farina E, Raglio A, Giovagnoli AR. Cognitive rehabilitation in epilepsy: An evidence-based review. Epilepsy Res. 2015 Jan;109:210-8. doi: 10.1016/j.eplepsyres.2014.10.017. Epub 2014 Nov 6. PMID 25524861
- [Background] Streltzov NA, Schmidt SS, Schommer LM, Zhao W, Tosteson TD, Mazanec MT, Kiriakopoulos ET, Chu F, Henninger HL, Nagle K, Roth RM, Jobst B. Effectiveness of a Self-Management Program to Improve Cognition and Quality of Life in Epilepsy: A Pragmatic, Randomized, Multicenter Trial. Neurology. 2022 May 24;98(21):e2174-e2184. doi: 10.1212/WNL.0000000000200346. Epub 2022 Apr 6. PMID 35387855
- [Background] Baxendale S. Cognitive rehabilitation and prehabilitation in people with epilepsy. Epilepsy Behav. 2020 May;106:107027. doi: 10.1016/j.yebeh.2020.107027. Epub 2020 Mar 21. PMID 32208338
- [Background] Rodakowski J, Saghafi E, Butters MA, Skidmore ER. Non-pharmacological interventions for adults with mild cognitive impairment and early stage dementia: An updated scoping review. Mol Aspects Med. 2015 Jun-Oct;43-44:38-53. doi: 10.1016/j.mam.2015.06.003. Epub 2015 Jun 10. PMID 26070444
- [Background] Daksla N, Nguyen V, Jin Z, Bergese SD. Brain Prehabilitation for Oncologic Surgery. Curr Oncol Rep. 2022 Nov;24(11):1513-1520. doi: 10.1007/s11912-022-01312-1. Epub 2022 Jul 28. PMID 35900715
- [Background] Humeidan ML, Reyes JC, Mavarez-Martinez A, Roeth C, Nguyen CM, Sheridan E, Zuleta-Alarcon A, Otey A, Abdel-Rasoul M, Bergese SD. Effect of Cognitive Prehabilitation on the Incidence of Postoperative Delirium Among Older Adults Undergoing Major Noncardiac Surgery: The Neurobics Randomized Clinical Trial. JAMA Surg. 2021 Feb 1;156(2):148-156. doi: 10.1001/jamasurg.2020.4371. PMID 33175114
- [Background] McCann M, Stamp N, Ngui A, Litton E. Cardiac Prehabilitation. J Cardiothorac Vasc Anesth. 2019 Aug;33(8):2255-2265. doi: 10.1053/j.jvca.2019.01.023. Epub 2019 Jan 12. PMID 30765210
- [Background] Smith NA, Martin G, Marginson B. Preoperative assessment and prehabilitation in patients with obesity undergoing non-bariatric surgery: A systematic review. J Clin Anesth. 2022 Jun;78:110676. doi: 10.1016/j.jclinane.2022.110676. Epub 2022 Feb 10. PMID 35152081
- [Background] Garcia-Delgado Y, Lopez-Madrazo-Hernandez MJ, Alvarado-Martel D, Miranda-Calderin G, Ugarte-Lopetegui A, Gonzalez-Medina RA, Hernandez-Lazaro A, Zamora G, Perez-Martin N, Sanchez-Hernandez RM, Ibarra-Gonzalez A, Bengoa-Dolon M, Mendoza-Vega CT, Appelvik-Gonzalez SM, Caballero-Diaz Y, Hernandez-Hernandez JR, Wagner AM. Prehabilitation for Bariatric Surgery: A Randomized, Controlled Trial Protocol and Pilot Study. Nutrients. 2021 Aug 24;13(9):2903. doi: 10.3390/nu13092903. PMID 34578781
- [Derived] Arrotta K, Babiker S, Lake J, Thompson N, Lioi A, Najm I, Busch RM. Readiness Brain Operation Optimization Training (ReBOOT) protocol: a feasibility randomised controlled trial for a cognitive prehabilitation programme for epilepsy surgery conducted at Cleveland Clinic, USA. BMJ Open. 2025 Nov 12;15(11):e091893. doi: 10.1136/bmjopen-2024-091893. PMID 41224310